CLINICAL TRIAL: NCT05156593
Title: 'Long COVID' in Suffolk and North Essex: Defining the Disease and Optimising Outcomes
Brief Title: 'Long COVID-19' in Suffolk and North Essex: Defining the Disease and Optimising Outcomes
Status: Completed | Type: Observational
Sponsor: East Suffolk and North Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20/187
Record Dates: First submitted 2021-12-09; First posted 2021-12-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2024-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To accurately describe the rehabilitation needs of individuals with post-COVID-19 syndrome up to 36 months after infection, allowing better diagnosis, triage and resource management. A major focus will be the impact on everyday life to return to normal activities.

ELIGIBILITY:
Inclusion criteria Individuals 18 years old and over (no upper age limit) Female and male Diagnosed with COVID-19 via PCR testing Or, Experienced symptoms of COVID-19 (new continuous cough, a high temperature, loss of taste and smell) And Clinically diagnosed with Post-COVID-19 Syndrome by their GP Participants who live within Suffolk and North East Essex

Exclusion criteria Individuals unable to consent for themselves Individuals without sufficient proficiency in English language to take part in telephone or video call, where the research team have been unable to make adjustments to enable their participation Individuals under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with diagnosed Long COVID
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Symptomology | 36 months
  Wide range of symptoms associated with Long COVID

CONTACTS AND LOCATIONS:
Overall Officials: Kate Harrall, Principal Investigator — East Suffolk and North Essex NHS Foundation Trust
Locations (1):
- East Suffolk and North Essex NHS Foundation Trust, Ipswich, United Kingdom